CLINICAL TRIAL: NCT04826406
Title: Camrelizumab Combined Apatinib in Patients With Hepatocellular Carcinoma Previously Treated With Immune Checkpoint Inhibitors: A Single-Arm, Open-Label, Phase II Study.
Brief Title: A Study of Camrelizumab Combined Apatinib in Hepatocellular Carcinoma Previously Treated With Immune Checkpoint Inhibitors (ICIs).
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Cancer Hospital (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-IIT-HCC
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Hepatocellular Carcinoma; Immune Checkpoint Inhibitors
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+Apatinib (Experimental)
  Interventions: Drug: Camrelizumab combined Apatinib regimen

INTERVENTIONS:
Drug: Camrelizumab combined Apatinib regimen — Camrelizumab 200mg iv every 2 weeks; Apatinib,250 mg/day.

SUMMARY:
The purpose of this study is to observe and preliminary explore the efficacy and safety of the combination of Camrelizumab and Apatinib regimen in treating advanced hepatocellular carcinoma (HCC) participants who have progressed following prior Immune Checkpoint Inhibitors (ICIs) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old, both genders.
* Conform to the clinical diagnosis histological or cytological confirmation of HCC(hepatocellular carcinoma) and with at least one measurable lesion by computed tomography (CT) scan or magnetic resonance imaging (MRI) according to RECIST 1.1.
* Liver function status Child-Pugh score less than or equal to 7.
* Barcelona Clinic Liver Cancer stage Category B or C.
* Disease progression following prior Immune Checkpoint Inhibitors (PD-1/PD-L1 or CTLA4 inhibitors) treatment for HCC, for at least 2 consecutive treatment cycles. Receipt of no more than 2 prior systemic therapies for advanced HCC.
* Eastern Cooperative Oncology Group Performance Status of 0 or 1.
* Life expectancy of at least 12 weeks.
* Adequate bone marrow, liver and renal function (without blood transfusion, without growth factor or blood components support within 14 days before enrollment).

Exclusion Criteria:

* Patients with any active autoimmune disease or history of autoimmune disease, including but not limited to the following: hepatitis, pneumonitis, uveitis, colitis (inflammatory bowel disease), hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Asthma that requires intermittent use of bronchodilators or other medical intervention should also be excluded.
* The prior ICIs treatments were discontinued by intolerable adverse events.
* Known or occurrence of central nervous system (CNS) metastases or hepatic encephalopathy.
* Patients with tumor burden ≥50% of the liver volume or received liver transplantation.
* Patients with clinical symptoms of ascites.
* Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents(within 3 months): systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg.
* Clinically significant cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, or coronary artery bypass surgery, Congestive heart failure (New York heart association (NYHA) class > 2), ventricular arrhythmia which need medical intervention.
* previous digestive tract bleeding history within 3 months or evident gastrointestinal bleeding tendency, such as: esophageal varices, local active ulcerative lesions, gastric ulcer and duodenal ulcer, the ulcerous colitis, gastrointestinal diseases such as portal hypertension or resection of tumor with bleeding risk, etc.
* Proteinuria ≥ (++) and 24 hours total urine protein > 1.0 g.
* Prior systemic chemotherapy, radiotherapy, immunotherapy, hormone therapy, surgery or target therapy within 4 weeks (or 5 half-life of the drug, calculate the longer ) before the study drug administration, or any unresolved AEs > Common Terminology Criteria for Adverse Events (CTCAE) Grade 1.
* Prior Camrelizumab or Apatinib treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2022-03-02 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 12 months
  Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Progression-free survival(PFS) | Up to approximately 12 months
  Progression-free survival(PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Time to objective response(TTR) | Up to approximately 12 months
  Time to objective response(TTR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Duration of Response (DoR) | Up to approximately 12 months
  Duration of Response (DoR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Disease Control Rate (DCR) | Up to approximately 12 months
  Disease Control Rate (DCR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
6-month survival rate | Up to approximately 12 months
  6-month survival rate
9-month survival rate | Up to approximately 12 months
  9-month survival rate
12-month survival rate | Up to approximately 12 months
  12-month survival rate
Overall survival(OS) | Up to approximately 24 months
Safety as measured by the rate of AEs, SAEs and laboratory abnormalities | From the first assignment of informed consent form up to 90 days after the last dose
  Safety as measured by the rate of AEs, SAEs and laboratory abnormalities (e.g. Grade 3 or higher per CTCAE v4 )

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided